CLINICAL TRIAL: NCT07312175
Title: A Study on 3D Printing-assisted Platelet-rich Plasma Combined With Autologous Periosteum-bone Grafting in the Treatment of Knee Cartilage Injury
Brief Title: 3D-Printed Grafts for Knee Cartilage Repair
Acronym: 3D-PR-PBG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-2025126
Record Dates: First submitted 2025-11-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Osteochondral Lesions of Knee; Osteo Arthritis
Keywords: Autologous osteoperiosteal transplantation; Massive; Osteochondral lesions; Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting (Experimental): 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting
  Interventions: Procedure: 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting; Procedure: 3D Printing-Assisted Autologous Periosteal-Bone Grafting
- 3D Printing-Assisted Autologous Periosteal-Bone Grafting (Other): 3D Printing-Assisted Autologous Periosteal-Bone Grafting
  Interventions: Procedure: 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting; Procedure: 3D Printing-Assisted Autologous Periosteal-Bone Grafting

INTERVENTIONS:
Procedure: 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting — 3D-Printed Scaffold-Assisted PRP Combined with Autologous Periosteal-Bone Grafting
Procedure: 3D Printing-Assisted Autologous Periosteal-Bone Grafting — 3D Printing-Assisted Autologous Periosteal-Bone Grafting

SUMMARY:
Research Title:A study on 3D printing-assisted platelet-rich plasma combined with autologous periosteum-bone grafting in the treatment of knee cartilage injury Objectives:(1) To evaluate the accuracy of cartilage damage repair by measuring the chimerism and surface curvature matching degree of 3D printing reconstruction. (2) 3D printing assisted platelerichplasma (PRP) combined with autologous periosteumBone grafting in patients with knee cartilage injury was evaluated for functional and imaging scores to evaluate the clinical effect and cartilage repair effect.

Design Type:Prospective randomized controlled trial Research Objects:Unilateral knee cartilage injury area>2CM2, international cartilagerepair society (ICRS) grade 3-4 patients Sample size: 60 cases (30 patients with 3D printing-assisted autologous periosteum-bone grafting, 3D printing-assisted PRP combined with autologous periosteum.) - 30 patients with bone grafting).Selection Criteria:(1) Age 18~65 years old; (2) The body mass index (BMI) is 18~30kg/m2 ； (3) Knee cartilage injury confirmed by imaging examination, knee cartilage injury 2>cm2, ICRS grade 3-4; (4) There is no obvious abnormality in the lower limb force line; (5) No other drug injection or surgical treatment has been performed locally in the knee joint in the past 1 year.

Observation indicators:(1) Clinical function(2) Imaging evaluation: Bilateral knee MRI examination was performed on the second day after surgery Statistical analysis methods:SPSS software was used for data analysis.

DETAILED DESCRIPTION:
Research Title:A study on 3D printing-assisted platelet-rich plasma combined with autologous periosteum-bone grafting in the treatment of knee cartilage injury Objectives:(1) To evaluate the accuracy of cartilage damage repair by measuring the chimerism and surface curvature matching degree of 3D printing reconstruction. (2) 3D printing assisted platelerichplasma (PRP) combined with autologous periosteumBone grafting in patients with knee cartilage injury was evaluated for functional and imaging scores to evaluate the clinical effect and cartilage repair effect.

Design Type:Prospective randomized controlled trial Research Objects:Unilateral knee cartilage injury area>2CM2, international cartilagerepair society (ICRS) grade 3-4 patients Sample size: 60 cases (30 patients with 3D printing-assisted autologous periosteum-bone grafting, 3D printing-assisted PRP combined with autologous periosteum.) - 30 patients with bone grafting).Selection Criteria:(1) Age 18~65 years old; (2) The body mass index (BMI) is 18~30kg/m2 ； (3) Knee cartilage injury confirmed by imaging examination, knee cartilage injury 2>cm2, ICRS grade 3-4; (4) There is no obvious abnormality in the lower limb force line; (5) No other drug injection or surgical treatment has been performed locally in the knee joint in the past 1 year.

Observation indicators:(1) Clinical function: Knee joint obtained by outpatient follow-up, written questionnaires, or by telephone by trained medical professionals before surgery and 1, 3, 6, and 12 months after surgery Lysholm score, Tegner exercise ability score, and pain numeric score were used to assess the improvement of symptoms and function. (2) Imaging evaluation: Bilateral knee MRI examination was performed on the second day after surgery, and the anatomical reconstruction was evaluated by mirror technology, including the chimerism of the bone bone interface between the graft and the host bone, and the match of the surface curvature of the graft and the recipient area. Magnetic resonanceobservationofcartilagerepairtissue observation (magneticresonanceobservationofcartilagerepairtissue, MOCART) scoring method scored MRI before surgery and 1 year after surgery to evaluate cartilage repair.

Statistical analysis methods:SPSS software was used for data analysis. The continuous data were expressed in (±s), and the normality test was performed, and the SNK test was used for comparison between groups. Repeated measures analysis of variance was used for comparison of time data before and after intervention within the group, and paired sample f test was used for comparison at two time points. If the data does not meet the normal distribution, the logarithmic transformation is analyzed again. The X2 test was used for the counting data. P<0.05 was a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. Body Mass Index (BMI) 18-30 kg/m²;
3. Imaging-confirmed knee cartilage damage >2 cm² with International Cartilage Repair Society (ICRS) grade 4;
4. No significant lower limb alignment abnormalities;
5. No prior local drug injections in the knee joint within the past year.

Exclusion Criteria:

1. Significant osteoporosis;
2. Individuals with immature bones;
3. Those with poor mechanical alignment;
4. Presence of meniscus injury, cruciate ligament or collateral ligament rupture, or incomplete healing following surgery for any of these conditions;
5. Severe knee joint effusion;
6. Use of corticosteroids or immunosuppressive agents;
7. Poor general health, alcoholism, or substance abuse;
8. Previous treatment with autologous blood products or stem cell preparations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical function | 1 year
  (1) Clinical function: Knee joint obtained by outpatient follow-up, written questionnaires, or by telephone by trained medical professionals before surgery and 1, 3, 6, and 12 months after surgery Lysholm score, Tegner exercise ability score, and pain numeric score were used to assess the improvement of symptoms and function.Lysholm score：minimum：0，maximum：80，a higher score represents a better outcome；Tegner exercise ability score：minimum：0，maximum：80，a higher score represents a better outcome；pain numeric score：minimum：0，maximum：10，a higher score represents a worse outcome.）

SECONDARY OUTCOMES:
Imaging evaluation | 1 year
  Imaging evaluation: Bilateral knee MRI examination was performed on the second day after surgery, and the anatomical reconstruction was evaluated by mirror technology, including the chimerism of the bone bone interface between the graft and the host bone, and the match of the surface curvature of the graft and the recipient area. Magnetic resonanceobservationofcartilagerepairtissue observation (magneticresonanceobservationofcartilagerepairtissue, MOCART) scoring method scored MRI before surgery and 1 year after surgery to evaluate cartilage repair.MOCART：minimum：0，maximum：10, a higher score represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- 330006, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-09-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT07312175/Prot_000.pdf